CLINICAL TRIAL: NCT00004483
Title: NF2 Natural History Consortium
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: House Ear Institute (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/14226; HEI-NF2; HEI-DAMD17-01-1-0710
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-09-29 (Estimated); Status verified 2005-09

CONDITIONS: Schwannoma, Vestibular; Neurofibromatosis 2; Meningioma
MeSH Terms: conditions — Neuroma, Acoustic; Neurofibromatosis 2; Meningioma

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

SUMMARY:
OBJECTIVES:

I. Define the growth rates and clinical course of NF2-related tumors in patients with neurofibromatosis type 2. Associate growth rate with physical function.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Data on the clinical course and growth rate of NF2-related tumors in patients with neurofibromatosis 2. Patients are evaluated each year on a cranial and a spinal MRI, eye tests, hearing tests, quality of life, neurological tests, and physical functioning.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnosed with neurofibromatosis 2 on or after 01/01/93
* Must meet one of the following conditions:

Bilateral vestibular schwannoma OR Family history of neurofibromatosis 2 (first degree family relative) AND Unilateral vestibular schwannoma at under 30 years OR Any 2 of the following: Meningioma Glioma Schwannoma Juvenile posterior subcapsular lenticular opacity/juvenile cortical cataract

* No plans to treat vestibular schwannoma in next 12 months

--Prior/Concurrent Therapy--

* Not specified

--Patient Characteristics--

* Age: 5 and over

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2002-01

CONTACTS AND LOCATIONS:
Overall Officials: William H. Slattery, III, Study Chair — House Ear Institute
Locations (1):
- House Ear Institute, Los Angeles, California, United States

REFERENCES:
- [Background] Masuda, Ann. Slattery, William H. III, Fisher, Laurel M., Oppenheimer, Mark. Audiological Characteristics of Initial Presentation of NF2 Patients: Preliminary Results. Abstract submitted to: Combined Otolaryngological Spring Meetings (COSM).
- [Background] Fisher, Laurel M., Slattery, WIlliam H. III, Yoon, Gloria. MRI Test-Retest Study of NF2 Patients. Abstract Submitted to: Combined Otolaryngological Spring Meetings (COSM).
- [Background] Slattery, William H. III, Fisher, Laurel M. Considerations in the Development of the NF2 Natural History Consortium. Submitted to Otolaryngology-Head and Neck Surgery.
- [Background] Masuda A, Fisher LM, Oppenheimer ML, Iqbal Z, Slattery WH; Natural History Consortium. Hearing changes after diagnosis in neurofibromatosis type 2. Otol Neurotol. 2004 Mar;25(2):150-4. doi: 10.1097/00129492-200403000-00012. PMID 15021775
- [Background] Slattery WH, Lev MH, Fisher LM, Connell SS, Iqbal Z, Go JL; NF2 Natural History Consortium. MRI evaluation of neurofibromatosis 2 patients: a standardized approach for accuracy in interpretation. Otol Neurotol. 2005 Jul;26(4):733-40. doi: 10.1097/01.mao.0000169048.15889.80. PMID 16015177
- [Background] Slattery WH 3rd, Fisher LM, Iqbal Z, Oppenhiemer M. Vestibular schwannoma growth rates in neurofibromatosis type 2 natural history consortium subjects. Otol Neurotol. 2004 Sep;25(5):811-7. doi: 10.1097/00129492-200409000-00027. PMID 15354016
- [Background] Zacharia, T., Lev, M., Iqbal, Z.T., Fisher ,L.M. , Gupta, MS, Slattery, WH. (2003) Intramedullary Spinal Tumors In NF II: Incidence And Imaging Characteristics American Radiology Society, 2003.